CLINICAL TRIAL: NCT03321929
Title: Feasibility Study Phase C: Expansion Into Multiple Institutions for Training in the Use of the LUM Imaging System for Intraoperative Detection of Residual Cancer in the Tumor Bed of Female Subjects With Breast Cancer
Brief Title: Intraoperative Detection of Residual Cancer in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumicell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL0006; 5R44CA211013-02 (NIH)
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LUM Imaging System (Experimental): Single dose of LUM015 (1.0 mg/kg) will be administered by intravenous injection between 2 to 6 hours prior to surgery. All subjects undergo lumpectomy as standard of care and will have the study intervention, guidance by intraoperative imaging using the LUM Imaging Device
  Interventions: Combination Product: LUM Imaging System

INTERVENTIONS:
Combination Product: LUM Imaging System — Drug: LUM015 Device: LUM 2.6 Imaging Device
  Other Names: LUM015

SUMMARY:
This is a non-randomized, open-label, multi-site study to collect safety and efficacy data on an intraoperative imaging system, the LUM Imaging System (LUM015 imaging agent in conjunction with the LUM imaging device), in identifying residual cancer in the tumor bed of female breast cancer patients. During the study, study physicians and clinical staff will complete hands-on training in anticipation of the upcoming pivotal study. Site-specific or user-specific issues related to the use of the device will be identified and addressed. Additionally, the data collected in the study will be used to continue training the tumor detection algorithm of the device.

In this study, patients will be injected with LUM015 prior to surgery. The study physicians will perform lumpectomy procedures according to his or her institution's standard of care practice. After the main specimen removal is completed, the study physician will use the LUM Imaging Device to image the tumor bed. Therapeutic shaves will be removed based on the recommendation of the LUM Imaging System. Patients will be followed until their first standard of care post-operative follow-up visit.

DETAILED DESCRIPTION:
For breast cancer lumpectomies, the presence of residual cancer cells left in the tumor bed after initial resection in inferred by post-operative margin assessment of the resected tissue by a pathologist.

Phase C enrollment will include approximately 5 patients per surgeon, with 2-3 surgeons per site and up to 20 sites. Subjects undergoing a lumpectomy procedure to treat primary breast cancer will be injected with a single dose of LUM015 4 ± 2 hours prior to surgery at a dose of 1.0 mg/kg. The sequence of events during the surgical procedure will vary based on the standard of care used by the surgeon. Patients will receive at a minimum the standard of care practices for each site. Lumicell-guided shaved cavity margins will be removed after the surgeon has attempted to remove the main specimen with grossly negative margins.

Study treatment ends when the surgery is completed. All patients will continue their enrollment in the study until their first follow-up visit and they will continue to be followed until the medical team determines no further surgical intervention is required. Patients with adverse events that are determined to be possibly related to the LUM Imaging System will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have histologically or cytologically confirmed primary invasive breast cancer, ductal carcinoma in situ (DCIS) or a combination of invasive breast cancer and DCIS. The protocol accepted methods for obtaining the histological samples are diagnostic core needle biopsies or fine needle biopsies.
* Female, age of 18 years or older. Because no dosing or adverse event data are currently available on the use of LUM015 in subjects <18 years of age, children are excluded from this study.
* Subjects must be scheduled for a lumpectomy for a breast malignancy.
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must have received and signed an informed consent form.
* Subjects must have no uncontrolled serious medical problems except for the diagnosis of cancer, as per the exclusion criteria listed below.
* Subjects must have normal organ and marrow function within limits as defined below:

  * Leukocytes > 3,000/mcL
  * Platelets > 75,000/mcL
  * total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine ≤ 1.5 mg/dL or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.

Exclusion criteria:

* Subjects who are treated for bilateral breast cancer resection procedure.
* Subjects who are pregnant at the time of diagnosis of their breast cancer; this exclusion is necessary because the teratogenic properties of LUM015 are unknown. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with LUM015, breastfeeding should be discontinued if the mother is treated with LUM015.
* Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception (hormonal or barrier method of birth control, abstinence) upon entering the study and for 60 days after injection of LUM015. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Breast cancer patients are routinely advised against becoming pregnant during treatment, so this requirement does not differ from standard of care.
* Subjects who have taken an investigational drug within 30 days of enrollment.
* Subjects with prolonged QTc interval defined as greater than 480 ms.
* Subjects who will have administration of methylene blue or any dye for sentinel lymph node mapping on the day of the surgery prior to imaging the lumpectomy cavity with the LUM Imaging Device.
* Subjects who have not recovered from adverse events due to other pharmaceutical or diagnostic agents.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 110 mm Hg; those subjects with known HTN should be stable within these ranges while under pharmaceutical therapy.
* History of allergic reaction attributed to drugs containing polyethylene glycol (PEG).
* History of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with LUM015.
* Any subject for whom the investigator feels participation is not in the best interest of the subject.
* Subjects undergoing a second lumpectomy procedure because of positive margins in a previous surgery prior to entering this study.
* Subjects with prior ipsilateral breast cancer surgeries, mastectomies, breast reconstructions or implants.
* Subjects who have undergone a surgical biopsy for any reason in the ipsilateral breast performed less than 2 years prior to enrollment of this study.
* Subjects with prior ipsilateral reduction mammoplasties (breast reductions) performed less than 2 years prior to enrollment to this study.
* Subjects previously treated with systemic therapies to treat the cancer to be removed during this clinical investigation, such as neo-adjuvant chemotherapy or hormonal therapy.
* Subjects undergoing breast conserving surgery whose resected specimen will be evaluated with frozen section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 234 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Smith, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (16):
- United States (16):
  - University of South Alabama, Mobile, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Comprehensive Breast Care Center, Clearwater, Florida
  - Baptist MD Anderson Cancer Physicians, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Beaumont Royal Oak, Royal Oak, Michigan
  - Beaumont Troy, Troy, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Dallas Breast Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Franciscan Breast Surgery, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang ES, Beitsch P, Blumencranz P, Carr D, Chagpar A, Clark L, Dekhne N, Dodge D, Dyess DL, Gold L, Grobmyer S, Hunt K, Karp S, Lesnikoski BA, Wapnir I, Smith BL; INSITE study team. Clinical Impact of Intraoperative Margin Assessment in Breast-Conserving Surgery With a Novel Pegulicianine Fluorescence-Guided System: A Nonrandomized Controlled Trial. JAMA Surg. 2022 Jul 1;157(7):573-580. doi: 10.1001/jamasurg.2022.1075. PMID 35544130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol, the enrolled population are those who were injected with LUM015.
Groups:
- LUM Imaging System: Single dose of LUM015 (1.0 mg/kg) will be administered by intravenous injection between 2 to 6 hours prior to surgery. All subjects undergo lumpectomy as standard of care and will have the study intervention, guidance by intraoperative imaging using the LUM Imaging Device
  LUM Imaging System: LUM015 will be administered 2 to 6 hours prior to surgery. All subjects will have intraoperative imaging using the LUM imaging device.
Period: Overall Study
Arm/Group | LUM Imaging System
Started | 234
Completed | 230 (Subjects withdrawn prior to LUM Imaging procedure completed were removed from the modified Intent to Treat population (mITT))
Not Completed | 4
Not completed — Withdrawn prior to LUM Imaging Procedure completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 220
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 187
  More than one race | 2
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 234
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] — Population: One patient did not have the height recorded in the system.
  Kg/m^2
    number analyzed (Participants) | 233
    (all) | 29.0 (6.6)
Menopausal Status [Count of Participants; unit: Participants]
  Post-menopausal | 187
  Pre/Peri-menopausal | 47
Mammographic breast density [Count of Participants; unit: Participants]
  Almost entirely fatty | 12
  Scattered areas of fibroglandular density | 119
  Heterogeneously dense | 86
  Extremely dense | 11
  Unknown | 6
Palpability [Count of Participants; unit: Participants]
  Palpable mass | 63
  Not palpable mass | 171

OUTCOME MEASURES:

1. Primary Outcome: Collect Data to Refine and Verify the Tumor Detection Algorithm.
Description: Data were collected from mITT population, which included all the patients imaged with the LUM Imaging System.
  This metric measured the residual cancer that current Standard of Care (SOC) lumpectomy failed to remove.
  It was defined as among all the patients, the percentage of subjects who had residual cancer found in at least one LUM-guided shave (therapeutic shave or "T-shave") after the current initial SOC lumpectomy procedure was completed.
Time Frame: 1 day
Population: modified intent to treat population (mITT) includes subjects injected with LUM015 and LUM Imaging was performed
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 230
Percentage | 11.3 [7.5 to 16.1]

2. Secondary Outcome: Number of Patients With Reported Adverse Events
Description: Reported adverse events will be assessed and aggregated according to event type, relation to device or drug, and severity.
Time Frame: Patients were evaluated for adverse events from time of injection until standard post-surgery follow-up visit (Median 31 days after lumpectomy).
Population: Subjects injected with LUM015 at a dose of 1mg/kg.
Measure: Count of Participants; unit: Participants
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 234
Participants
  Chromaturia Adverse Events: number analyzed (Participants) | 214
  Chromaturia Adverse Events: Mild or Moderate, Not Related | 0
  Chromaturia Adverse Events: Mild or Moderate, Related | 214
  Chromaturia Adverse Events: Severe, Not Related | 0
  Chromaturia Adverse Events: Severe, Related | 0
  Chromaturia Adverse Events: Life Threatening, Not Related | 0
  Chromaturia Adverse Events: Life Threatening, Related | 0
  Non Chromaturia Adverse Events: number analyzed (Participants) | 36
  Non Chromaturia Adverse Events: Mild or Moderate, Not Related | 33
  Non Chromaturia Adverse Events: Mild or Moderate, Related | 1
  Non Chromaturia Adverse Events: Severe, Not Related | 0
  Non Chromaturia Adverse Events: Severe, Related | 1
  Non Chromaturia Adverse Events: Life Threatening, Not Related | 0
  Non Chromaturia Adverse Events: Life Threatening, Related | 1

3. Secondary Outcome: Tumor Removal Rate in the Whole mITT Population by SOC Margin Status
Description: Collect data to verify the detection algorithm reported in previous studies by SOC margin status
Time Frame: 1 week
Measure: Number (95% Confidence Interval); unit: Percentage of All Subjects
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 230
Percentage of All Subjects
  Percentage of subjects with positive SOC margins having tumor in at least one therapeutic shave. | 5.2 [2.7 to 8.9]
  Percentage of subjects with negative SOC margins having tumor in at least one therapeutic shave. | 6.1 [3.4 to 10.0]

4. Secondary Outcome: Tumor Removal Rate Within Subjects Having Positive Standard of Care Margins
Description: Tumor removal rate was measured as the percentage of the subjects who had residual tumor removed guided by Lumicell Imaging System after standard of care (SOC) procedure within subjects who had positive margins after SOC.
Time Frame: 1 Week
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 38
Percentage of Subjects | 31.6 [17.5 to 48.7]

5. Secondary Outcome: Tumor Removal Rate Within Subjects Having All Negative SOC Margins
Description: Tumor removal rate was measured as the percentage of the subjects who had residual tumor removed guided by Lumicell Imaging System after standard of care (SOC) procedure within subjects who had negative margins after SOC.
Time Frame: 1 Week
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 192
Percentage of Subjects | 7.3 [4 to 11.9]

6. Secondary Outcome: Sensitivity and Specificity of the LUM Imaging System in Predicting Residual Cancer in the Cavity
Description: Sensitivity and specificity were measured at the tissue level for the Lumicell imaging signal for the sensitivity and specificity on the residual tumor in the cavity of corresponding orientations after standard of care (SOC) of Lumpectomy. Generalized Estimating Equation (GEE) has been applied using generalized linear model having binomial link function and compound symmetry working correlation structure within each subject.
Time Frame: 1 Week
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 230
Percentage
  Sensitivity (GEE) | 69.3 [55.8 to 80.1]
  Specificity (GEE) | 71.7 [68.5 to 74.7]

7. Secondary Outcome: Detection and Conversion of Positive Margins in Subjects After BCS SOC
Description: Conversion was measured as the ratio of the subjects having all the positive margins after BCS SOC converted to negatives after Lumicell Imaging guided procedure.
  Detection was measured as the ratio of the subjects having all or at least one positive margin after BCS SOC detected by Lumicell Imaging System.
  BCS: Breast-conserving surgery; SOC: Standard of Care
Time Frame: 1 Week
Measure: Number (95% Confidence Interval); unit: Percentage of All Subjects
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 38
Percentage of All Subjects
  Percentage of Subjects Having SOC Positive Margins All Converted to Negative | 15.8 [6 to 31.3]
  Percentage of Subjects Having SOC Positive Margins All Detected by Lumicell Device | 28.9 [15.4 to 45.9]
  Percentage of Subjects Having At Least One SOC Positive Margin Detected by Lumicell Device | 42.1 [26.3 to 59.2]

8. Secondary Outcome: Volume of Therapeutic Shaves Removed During Lumpectomy.
Description: The median volumes of Lumicell Imaging System - guided shaves (therapeutic shaves) were measured and the median total volume removed during lumpectomy was presented as well.
Time Frame: 1 Week
Population: Total mITT population
Measure: Median (95% Confidence Interval); unit: Volume in CM^3
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 230
Volume in CM^3
  Lumpectomy volume (cm3) | 57.8 [11.5 to 252.7]
  SOC shave volume (cm3) | 6.0 [0.0 to 52.5]
  SOC total volume (cm3) | 65.4 [17.9 to 276.9]
  Therapeutic shave volume (cm3) | 4.0 [0.0 to 102.8]
  Total volume (cm3) | 77.7 [18.8 to 336.8]

9. Other Pre Specified Outcome: Number of Surgeons Trained on the Use of the LUM Imaging System
Description: Surgeons were trained on using the LUM Imaging System in preparation for participating in future clinical trials with the LUM Imaging System. Workflows were established at each institution to support the use of the LUM Imaging System and protocol adherence during lumpectomy procedures. Surgeons were not participants in the trial. Surgeons were the Investigators in the trial.
Time Frame: 1 day
Population: Thirty-eight surgeons at 16 clinical sites were trained on the use of the LUM Imaging System.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Surgeons Trained on Using the LUM Imaging System: Surgeons were trained on using the LUM Imaging System in preparation for participating in future clinical trials with the LUM Imaging System. Workflows were established at each institution to support the use of the LUM Imaging System and protocol adherence during lumpectomy procedures. Surgeons were not participants in the trial.
Arm/Group | Number of Surgeons Trained on Using the LUM Imaging System
Number analyzed (Participants) | 38
Participants | 38

10. Secondary Outcome: Contribution of Therapeutic Shaves to Total Volume Removed During Lumpectomy.
Description: The contribution of the volumes of Lumicell Imaging System - guided shaves (therapeutic shaves) were measured as percentage of the sum of the volumes of the therapeutic shaves out of the total volume removed during lumpectomy.
Time Frame: 1 Week
Population: Total mITT population
Measure: Median (95% Confidence Interval); unit: Percentage
Arm/Group | LUM Imaging System
Number analyzed (Participants) | 230
Percentage | 6.5 [0 to 55.9]

ADVERSE EVENTS:
Time Frame: All adverse events and adverse device effects, both serious and non-serious, and deaths that are encountered from initiation of study intervention, throughout the study, and within the first post-operative follow-up visit should be followed to their resolution, or until the principal investigator assesses them as stable, or the principal investigator determines the event to be irreversible, or the subject is lost to follow-up. Adverse events were assessed up to 30 days after enrollment.
Description: Serious adverse events should be reported within 24 hours of learning of the occurrence. Non-serious adverse events and non-serious adverse device effects will be reported to Lumicell on the adverse events Case Report Forms during the study.
Arm/Group | LUM Imaging System
All-Cause Mortality (participants affected / at risk) | 0/234
Serious Adverse Events (participants affected / at risk) | 1/234
Other Adverse Events (participants affected / at risk) | 215/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM Imaging System (N=234)
Anaphylactic Reaction (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than .9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM Imaging System (N=234)
Chromaturia (Renal and urinary disorders) | 214 (214)
Seroma (Injury, poisoning and procedural complications) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)

LIMITATIONS AND CAVEATS:
Protocol deviations may have impacted the reported performance. In some patients no LUM shaves were removed either because of protocol deviation or because the protocol limited the number of additional shaves that could be excised at any single margin. These deviations may have precluded full pathologic correlation and evaluation of clinical utility for many of the LUM images and may have prevented conversion of positive margins to negative margins.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03321929/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT03321929/SAP_001.pdf